CLINICAL TRIAL: NCT05589974
Title: Choroidal Blood Flow in Acute and Chronic Central Serous Chorioretinopathy
Status: Recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: REK485079
Record Dates: First submitted 2022-09-20; First posted 2022-10-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-11

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Verteporfin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute: Patients with acute first attack CSC with subretinal fluid (SRF) on OCT and symptom duration under 4 months.
- Chronic: Patients with chronic CSC, i.e. symptoms and SRF for more than 4 months.
  Interventions: Drug: Verteporfin

INTERVENTIONS:
Drug: Verteporfin — Chronic CSC are receiving one treatment before the observation period.
  Groups: Chronic

SUMMARY:
Patients with central serous chorioretinopathy (CSC) will be monitored with laser speckle flow graphy (LSFG), swept source optical coherence tomography (SS-OCT) and SS-OCT angiography (SS-OCTA). The aim is to unveil the flow and pulse wave characteristics of the choroidal circulation in acute CSC and chronic CSC.

DETAILED DESCRIPTION:
Acute CSC - The proposed study tests the hypothesis that choroidal blood flow characteristics are related to the eventual resolution of subretinal fluid. Such relation can shed light on pathophysiological disease mechanisms and constitute a biomarker for disease activity.

Chronic CSC - The proposed study tests the hypothesis that choroidal blood flow characteristics will change in response to standard treatment with PDT. The research of such changes will increase the understanding of the treatment response. This knowledge will help in the effort to understand the why some patients are non-responsive to the treatment.

ELIGIBILITY:
Inclusion Criteria:-

* Able to sign informed consent
* Possible to obtain fundus imaging
* Acute CSC ˂4 months of duration in one eye, defined as:

  1. Subfoveal presence of SRF on OCT
  2. Present attack is 1st -3rd attack of CSC

  b) Patient history and examination consistent with acute CSC c) Characteristic appearance of acute CSC on fundus autofluorescence (FAF) and OCT
* Chronic CSC ≥4 months of duration in one eye, defined as:

  1. Subfoveal presence of SRF on OCT
  2. Subjective visual loss/symptoms
  3. Characteristic appearance of chronic CSC on FAF, fluorescein angiography (FA), and indocyanin angiography (ICGA) and OCT
  4. Patient history and examination consistent with chronic CSC

Exclusion Criteria:

* History of retinal disease other than CSC (e.g. retinal detachment)
* Contraindications for FA, ICGA or PDT (only for chronic CSC)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute or chronic CSC.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean blur rate | 6 months
  Relative changes in choroidal blood flow
Change in pulse wave form analysis | 6 months
  Changes in the shapes of pulse curves

SECONDARY OUTCOMES:
Change in choroidal density | 6 months
  Changes in the tissue density
Change in choroidal thickness | 6 months
  Changes in the morphology of the choroid

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Forsaa, MD PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Department of Ophthalmology, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: Yes
This study can be expanded as a multicenterstudy. I so, IPD will be shared among the study group.
Supporting Information: Study Protocol, SAP, ICF, CSR